CLINICAL TRIAL: NCT00114387
Title: VEAPS: Vitamin E Atherosclerosis Prevention Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AG0023; R01AG013860 (NIH)
Record Dates: First submitted 2005-06-14; First posted 2005-06-15 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2005-06

CONDITIONS: Atherosclerosis
Keywords: vitamin E
MeSH Terms: conditions — Atherosclerosis | interventions — alpha-Tocopherol

INTERVENTIONS:
Drug: DL-alpha-tocopherol

SUMMARY:
The purpose of this study is to examine whether vitamin E (DL-alpha-tocopherol) supplementation will reduce the progression of early atherosclerosis in healthy individuals over 40 years of age with low-density lipoprotein (LDL) cholesterol levels greater than or equal to 130mg/dL.

DETAILED DESCRIPTION:
The primary hypothesis to be tested is that vitamin E supplementation of 400 IU/day exerts positive arterial wall effects by reducing progression of early atherosclerosis in healthy individuals 40 years old or older without clinical evidence of cardiovascular disease (CVD). Ultrasonography will be used to measure the rate of change of the distal common carotid artery (CCA) far wall intima-media thickness (IMT). The beneficial effects of vitamin E supplementation are expected to occur with or without a change in LDL-C levels.

A total of 353 men and women will be recruited for the three-year trial. Participants will be randomized into a treatment group to receive either vitamin E (DL-alpha-tocopherol) 400 IU/day or a placebo. The ultrasound measurement of CCA IMT will be repeated every six months for two years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 40 years or older
* Fasting LDL-C level 130 mg/dL or greater, TG (triglyceride) levels 500mg/dL or lower

Exclusion Criteria:

* Any clinical signs or symptoms of cardiovascular disease (CVD)
* Diabetes mellitus or fasting serum glucose 140mg/dL or greater
* Regular vitamin E supplementation for more than 1 year
* Lipid standardized plasma vitamin E levels greater than 35 micromoles per liter (μmol/L)
* Uncontrolled hypertension (diastolic blood pressure 100 mmHg or greater)
* Thyroid disease (untreated)
* Renal insufficiency (serum creatinine greater than 2.5 mg/dL)
* Life threatening disease with prognosis less than 5 years
* Alcohol intake greater than 5 drinks per day (1 drink = 1 1/2 oz distilled spirits, 4 oz wine, or 12 oz beer) or substance abuse (intravenous drug abuse, cocaine use)

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 353
Dates: Start 1996-07; Primary Completion 2000-09 (Actual); Study Completion 2000-09 (Actual)

PRIMARY OUTCOMES:
Rate of change of the distal common carotid artery (CCA) far wall intima-media thickness (IMT)

CONTACTS AND LOCATIONS:
Overall Officials: Howard N. Hodis, MD, Principal Investigator — University of Southern California, Atherosclerosis Research Unit, Division of Cardiovascular Medicine, Department of Medicine
Locations (1):
- Atherosclerosis Research Unit, Division of Cardiovascular Medicine, Department of Medicine, Los Angeles, California, United States

REFERENCES:
- [Result] Hodis HN, Mack WJ, LaBree L, Mahrer PR, Sevanian A, Liu CR, Liu CH, Hwang J, Selzer RH, Azen SP; VEAPS Research Group. Alpha-tocopherol supplementation in healthy individuals reduces low-density lipoprotein oxidation but not atherosclerosis: the Vitamin E Atherosclerosis Prevention Study (VEAPS). Circulation. 2002 Sep 17;106(12):1453-9. doi: 10.1161/01.cir.0000029092.99946.08. PMID 12234947
- [Derived] Huang J, Hodis HN, Weinstein SJ, Mack WJ, Sampson JN, Mondul AM, Albanes D. Serum Metabolomic Response to Low- and High-Dose Vitamin E Supplementation in Two Randomized Controlled Trials. Cancer Epidemiol Biomarkers Prev. 2020 Jul;29(7):1329-1334. doi: 10.1158/1055-9965.EPI-20-0187. Epub 2020 Apr 20. PMID 32312759